CLINICAL TRIAL: NCT05963295
Title: Toxoplasma Gondii Infection in Both Children and Adult Patients With Hematological Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Norhan Mohamed Abdelhalim, resident-clinical pathology sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-23-07-16MS
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient with hematlolgical malignancies (Active Comparator)
  Interventions: Diagnostic Test: toxoplasma igG
- control group (Active Comparator)
  Interventions: Diagnostic Test: toxoplasma igG

INTERVENTIONS:
Diagnostic Test: toxoplasma igG — Dignosis of toxoplasma
  Other Names: toxoplasma IgM

SUMMARY:
Toxoplasmosis is one of the most common zoonotic diseases caused by the obligate intracellular parasite, T. gondii. It affects up to one-third of the world's population Horizontal transmission is mostly caused by ingestion of tissue cysts in infected meat, or through consumption of food or drink contaminated with sporulated oocysts, while vertical transmission occurs due to primary acquired maternal infection throughout pregnancy.In immunocompetent hosts, acquired infection is asymptomatic in more than 80% of cases, or is associated with fever,cervical lymphadenopathy, or myalgia.

In immunocompromised patients,toxoplasmosis is always life-threatening where toxoplasmic encephalitis is the most important presentation. Among those patients, the disease may be caused by a newly acquired infection, reactivation following cyst rupture, donation of a cyst-containing organ from a seropositive donor to a seronegative recipient, or reactivation of dormant infection in the recipient Patients with hematological malignancy (HM), including those with acute myelogenous leukemia, and those who have undergone hematopoietic stem cell transplantation or treated with aggressive immunosuppressive regimens are at high risk of opportunistic infections The association between toxoplasmosis and cancers remains dual. Most cancer patients are in a state of impaired cellular and humoral immune systems either from the primary disease, or from chemotherapy and/or radiotherapy administration. Chemotherapeutic drugs work by killing both fast growing cancer cells, and healthy white blood cells causing neutropenia. So, patients receiving chemotherapy are more susceptible to Toxoplasma infections.

Many studies have reported that the rate of reactivation of a latent T. gondii infection was higher in different types of cancers particularly those of the eye, brain, blood and breast. On the other side, T. gondii was also implicated as possible oncogenic pathogen with suggested role in induction and progression of malignant diseases. This was explained by many theories such as preventing apoptosis, enhancing the motility of dendritic cells and macrophages.

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted on a group of patients who are diagnosed as have hematological malignancies

Exclusion Criteria:

* Patients with other non hematological malignancies.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
toxoplasma IgG | 1 year
  rising titre

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elzeny H, Mohamed W, Daef E, El-Badawy O, Shaaban L, Osman NS, Hadiya S, Aly S. Detection of multiple extensively-drug resistant hypervirulent Klebsiella pneumoniae clones from patients with ventilator-associated pneumonia in Egypt. J Med Microbiol. 2023 Jun;72(6). doi: 10.1099/jmm.0.001701. PMID 37288576
- [Background] Dupont D, Fricker-Hidalgo H, Brenier-Pinchart MP, Garnaud C, Wallon M, Pelloux H. Serology for Toxoplasma in Immunocompromised Patients: Still Useful? Trends Parasitol. 2021 Mar;37(3):205-213. doi: 10.1016/j.pt.2020.09.006. Epub 2020 Oct 9. PMID 33046380
- [Background] Anvari D, Sharif M, Sarvi S, Aghayan SA, Gholami S, Pagheh AS, Hosseini SA, Saberi R, Chegeni TN, Hosseininejad Z, Daryani A. Seroprevalence of Toxoplasma gondii infection in cancer patients: A systematic review and meta-analysis. Microb Pathog. 2019 Apr;129:30-42. doi: 10.1016/j.micpath.2019.01.040. Epub 2019 Jan 29. PMID 30708042
- [Background] Kalantari N, Gorgani-Firouzjaee T, Hassani S, Chehrazi M, Ghaffari S. Association between Toxoplasma gondii exposure and hematological malignancies: A systematic review and meta-analysis. Microb Pathog. 2020 Nov;148:104440. doi: 10.1016/j.micpath.2020.104440. Epub 2020 Aug 19. PMID 32822769